CLINICAL TRIAL: NCT03266653
Title: A Pilot Study in the Treatment of Refractory Epstein-Barr Virus (EBV) Infection With Related Donor EBV Cytotoxic T-Lymphocytes in Children, Adolescents and Young Adult Recipients
Brief Title: EBV-specific Cytotoxic T-lymphocytes (CTLs) for Refractory EBV Infection
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: New York Medical College (Other)
Collaborators: Children's Hospital of Philadelphia (Other); Medical College of Wisconsin (Other); Nationwide Children's Hospital (Other); Indiana University (Other); Washington University School of Medicine (Other); University of California, Los Angeles (Other); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Mitchell Cairo, Principal Investigator, New York Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYMC 581; FD006363 (Other Grant/Funding Number: FDA OOPD)
Record Dates: First submitted 2017-08-25; First posted 2017-08-30 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Epstein-Barr Virus Infections; Primary Immune Deficiency Disorder
MeSH Terms: conditions — Epstein-Barr Virus Infections; Primary Immunodeficiency Diseases

STUDY DESIGN:
Intervention Model Description: All patients given identical treatment with CTLs for refractory EBV.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Refractory EBV (Experimental): Patients with refractory EBV will get one dose of EBV specific CTLs. If they don't show a response based on EBV PCRs, patients may get up to another 4 doses of EBV-CTLs (5 doses maximum)
  Interventions: Drug: cytotoxic t-lymphocytes

INTERVENTIONS:
Drug: cytotoxic t-lymphocytes — EBV specific CTLs will be generated from HLA related matched and mismatched donors in a GMP facility and administered to the patient with refractory CTLs.
  Other Names: CTLs

SUMMARY:
Related donor Epstein-Barr Virus (EBV) specific cytotoxic T cells (CTLs) manufactured with the Miltenyi CliniMACS Prodigy Cytokine Capture System will be administered in children, adolescents and young adults with refractory EBV infection post Allogeneic Hematopoietic Stem Cell Transplantation (AlloHSCT), with primary immunodeficiencies (PID) or post solid organ transplant.

Funding Source: FDA OOPD

ELIGIBILITY:
1. Patients with Epstein-Barr virus infections post allogeneic HSCT, primary immunodeficiencies or post solid organ transplant with:

* Increasing or persistent quantitative EBV RT-PCR DNA copies despite two weeks of appropriate anti-viral therapy and/or
* progressive clinical symptoms attributable to EBV, including biopsy proven colitis, lymphadenopathy, hepatomegaly, splenomegaly AND/OR
* Medical intolerance to anti-viral therapies including:
* intolerance to rituximab Consent: Written informed consent given (by patient or legal representative) prior to any study-related procedures.

Performance Status > 30% (Lansky < 16 yrs and Karnofsky > 16 yrs) Age: 0.1 to 79.99 years Females of childbearing potential with a negative urine pregnancy test

2 Donor Eligibility 5.2.1 Related donor available with a T-cell response to the EBV MACS® GMP PepTivator antigen(s) causing the therapy-refractory EBV infection.

a. Third Party Related Allogeneic Donor: If original donor is not available or does not have a T-cell response: third party related allogeneic donor (family donor > 1 HLA A, B, DR match to recipient) with IgG positive to EBV and/or a T-cell response at least to the viral MACS® GMP PepTivator EBV Select (containing among other antigens, NA-1, LMP2A and BZLF-1).

AND Allogeneic donor disease screening is complete similar to hematopoietic stem cell donors (Appendix 1).

AND Obtained informed consents by donor or donor legally authorized representative prior to donor collection.

3 Patient exclusion criteria:

A patient meeting any of the following criteria is not eligible for the present study:

Patient with acute GVHD > grade 2 or extensive chronic GVHD at the time of CTL infusion Patient receiving steroids (>0.5 mg/kg prednisone equivalent) at the time of CTL infusion Patient treated with donor lymphocyte infusion (DLI) within 4 weeks prior to CTL infusion Patient with poor performance status determined by Karnofsky (patients >16 years) or Lansky (patients ≤16 years) score ≤30% Concomitant enrollment in another experimental clinical trial investigating the treatment of refractory EBV infection Any medical condition which could compromise participation in the study according to the investigator's assessment Known HIV infection Female patient of childbearing age who is pregnant or breast-feeding or not willing to use an effective method of birth control during study treatment.

Known hypersensitivity to iron dextran Patients unwilling or unable to comply with the protocol or unable to give informed consent.

Known human anti-mouse antibodies

Ages: 1 Month to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-07-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Patients will be followed for 12 weeks after each infusion
  Patients will be monitored for adverse events related to the infusion of EBV CTLs
Incidence of Response to Treatment [Efficacy] | Patients will be followed for 12 weeks after each infusion
  Patients will be followed for improvement in viral infection by monitoring EBV PCR weekly for response to treatment with CTLs

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Cairo, MD, Principal Investigator — New York Medical College
Locations (8):
- United States (8):
  - Children's Hosptial Los Angeles, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Johns Hopkins, Baltimore, Maryland
  - Washington University, St Louis, Missouri
  - New York Medical College, Valhalla, New York
  - Nationwide Children's Hosptial, Columbus, Ohio
  - Children's Hospital of Pennsylvania, Philadelphia, Pennsylvania
  - Medical College of Wisconsin/Children's Hospital of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided